CLINICAL TRIAL: NCT06366893
Title: Enteral Supplementation With Docosahexaenoic Acid and Arachidonic Acid (DHA-AA) in Preterm Infants. Single-center, Prospective, Randomized, Controlled, Open-label Clinical Trial
Brief Title: Enteral Supplementation With Docosahexaenoic Acid and Arachidonic Acid (DHA-AA) in Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR(AG)297/2019
Record Dates: First submitted 2024-01-31; First posted 2024-04-16 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Infant, Premature, Diseases
Keywords: docosahexaenoic acid; arachidonic acid; erythrocyte membrane; preterm infants; supplementation
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The study group will be supplemented with DHA and AA emulsion for 28 days. Patients will be followed up until hospital discharge. The emulsion will be administered by nasogastric or orogastric tube together with the scheduled milk intake (from the bank or the mother's own with a differentiated amount of supplementation depending on the type of milk administered and the infant's weight).
  Interventions: Dietary Supplement: DHA/AA emulsion supplement for preterm infant
- Control group (No Intervention): The control group will not be supplemented with DHA and AA emulsion. Patients will be followed up until hospital discharge.

INTERVENTIONS:
Dietary Supplement: DHA/AA emulsion supplement for preterm infant — Enteral supplementation of DHA/AA emulsion
  Arms: Study group

SUMMARY:
Docosahexaenoic acid (DHA) and arachidonic acid (AA) have a critical effect on the health and neuronal development of the fetus and newborn. Their deficiency has been associated with increased neonatal morbidity, especially in preterm newborns at birth. Direct DHA supplementation during the first few weeks of life could prevent this deficiency.

The aim is to increase DHA levels in the red blood cell membrane while maintaining the fetal proportion to AA in preterm infants through enteral administration of DHA/AA in a safe, tolerated, and effective manner. This approach aims to avoid the decline in DHA/AA levels and the consequences of their deficiency.

The study is a single-center, prospective, randomized, controlled, open-label study involving preterm infants admitted to the Neonatology Department of Vall d'Hebron University Hospital in Barcelona.

DETAILED DESCRIPTION:
Polyunsaturated fatty acids (PUFAs), especially DHA and AA, are essential fatty acids that have a high relevance in the growth and development of the fetus and newborn. Preterm infants are at high risk of suffering from a deficiency of these essential fatty acids. This deficit would cause serious visual impairments and alterations in neuronal development, as well as an increase in morbidity in these patients.

The external contribution after birth is mainly based on that provided through the mother's own milk (premature milk) and when it is not sufficient, it is supplemented with bank milk. This enteral milk intake is not complete until after the first week of life. In addition, the proportion of bank milk administered in this phase is higher than the mother's own milk. This bank milk has a lower concentration of DHA mainly.

If complete enteral feeding is not achieved until 10 days of age and this is mainly done at the expense of bank milk with a lower DHA content than the mother's premature milk, it seems reasonable to directly supplement the preterm infant with DHA and AA from the first days of life as indicated with other fortifications and thus avoid the risk of deficiency and its consequences. This intake should be similar to that of assimilated intrauterine: 50-60 mg/kg/day. Despite these statements, specific and direct supplementation of DHA and AA is not carried out as standard clinical practice in preterm infants. They have only been carried out in the context of studies.

Enteral supplementation of DHA and AA during the first month of life in the preterm newborn will ensure optimal levels of DHA and AA similar to those achieved in intrauterine life, which will be essential for the correct growth of the newborn and its optimal neuronal development.

This supplementation is not a common healthcare practice in the Neonatology Departments. Our study proposes a safe and effective way to avoid DHA and AA deficiency in the first days of life and its consequences.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with a gestational age between 23 and 32 weeks admitted to the Neonatology Service of the Vall d'Hebron University Hospital and with informed consent signed by the parents or legal guardians.

Exclusion Criteria:

* Severe malformation incompatible with life.
* Impossibility of enteral nutrition during the expected duration of the study (30 days).

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-03-04 (Estimated); Study Completion 2025-03-04 (Estimated)

PRIMARY OUTCOMES:
Percentage comparison of erythrocyte membrane levels of DHA and AA | 4 weeks
  Compare the percentage erythrocyte membrane levels of DHA and AA during the first month of life between the supplemented group and the control group.

SECONDARY OUTCOMES:
Tolerance of DHA emulsion administration | 4 weeks
  Number of days when enteral nutrition prescriptions have had to be suspended.
Compare the presence of pathologies in preterm infants between the supplemented group and the control group | 4 weeks
  Tracking data related to:
  * Bronchopulmonary dysplasia (BPD)
  * Retinopathy of prematurity (ROP)
  * Sepsis
  * Necrotizing enterocolitis:
  * Intraventricular hemorrhage and periventricular leukomalacia

CONTACTS AND LOCATIONS:
Overall Officials: Félix Castillo Salinas, Dr., Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Materno Infantil Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castillo Salinas F, Montaner Ramon A, Castillo Ferrer FJ, Domingo-Carnice A, Cordobilla B, Domingo JC. Erythrocyte Membrane Docosahexaenoic Acid (DHA) and Lipid Profile in Preterm Infants at Birth and Over the First Month of Life: A Comparative Study with Infants at Term. Nutrients. 2022 Nov 22;14(23):4956. doi: 10.3390/nu14234956. PMID 36500985
- [Background] Castillo F, Castillo-Ferrer FJ, Cordobilla B, Domingo JC. Inadequate Content of Docosahexaenoic Acid (DHA) of Donor Human Milk for Feeding Preterm Infants: A Comparison with Mother's Own Milk at Different Stages of Lactation. Nutrients. 2021 Apr 15;13(4):1300. doi: 10.3390/nu13041300. PMID 33920807